CLINICAL TRIAL: NCT07358572
Title: A Study on the Eye-Brain-Kidney Interaction Mechanisms in Chronic Kidney Disease Based on Multimodal Magnetic Resonance Imaging
Brief Title: Eye-Brain-Kidney in CKD
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EBK-CKD
Record Dates: First submitted 2025-12-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Multimodal magnetic resonance imaging; Montreal Cognitive Assessment
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum and plasma samples obtained from the remaining blood after routine complete blood count and biochemistry tests. These samples will be stored in a biobank for centralized analysis of disease-related biomarkers, including but not limited to Tau, phosphorylated Tau, phenylacetylglutamine, indole acetic acid, and β2-microglobulin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the interaction between the eyes, brain, and kidneys in adult patients with Chronic Kidney Disease (CKD). The main question it aims to answer is:

Do changes in the brain's network connectivity and the retina's blood vessels correlate with cognitive decline and kidney function in CKD patients? Participants with CKD who are already undergoing clinical care will complete cognitive tests and questionnaires, have non-invasive MRI scans of their brain and kidneys, and undergo non-invasive eye imaging (OCT/OCTA) of their retinas.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational cohort study designed to investigate the multi-system interactions among the eyes, brain, and kidneys in patients with Chronic Kidney Disease (CKD) stages 1-5. The study integrates multimodal imaging, clinical laboratory tests, and neuropsychological assessments to establish a comprehensive "eye-brain-kidney" evaluation framework.

Study Design and Procedures:

The study plans to enroll CKD patients from Beijing Friendship Hospital, Capital Medical University, between December 2025 and December 2028. All enrolled participants will undergo comprehensive evaluations at two time points: baseline and a 3-year follow-up. Baseline assessments include: medical history collection, neuropsychological scale evaluations (Montreal Cognitive Assessment, Symbol-Digit Modalities Test, Digit Span Test, Hospital Anxiety and Depression Scale), blood tests (complete blood count, biochemistry, and specific biomarkers such as Tau protein and β2-microglobulin), multimodal brain magnetic resonance imaging (MRI), multiparametric kidney MRI, and ocular optical coherence tomography (OCT). The above assessments will be repeated at the 3-year follow-up to observe longitudinal changes in all parameters.

Assessment Methods and Technical Parameters:

1. Brain MRI: A 3.0T MRI scanner will be used to acquire multiple sequences including 3D T1-weighted structural imaging, resting-state functional MRI, arterial spin labeling perfusion imaging, diffusion tensor imaging, quantitative susceptibility mapping, and amide proton transfer-chemical exchange saturation transfer imaging. These will be used to analyze brain structure, perfusion, functional connectivity, and metabolic changes.
2. Kidney MRI: A 3.0T MRI scanner will be used with sequences such as intravoxel incoherent motion, arterial spin labeling, and T1 mapping to quantitatively assess renal microcirculation perfusion, tissue diffusion characteristics, and the degree of fibrosis.
3. Ocular Imaging: Optical coherence tomography and angiography will be used to obtain quantitative parameters including retinal nerve fiber layer thickness, macular structure, choroidal thickness, and vessel density in the superficial and deep retinal capillary plexuses.
4. Clinical and Cognitive Assessments: In addition to standardized scales, remaining serum and plasma samples from participants will be preserved for subsequent biomarker analysis.

Quality Control and Data Management:

A comprehensive quality control plan has been developed and implemented for this study:

Data Acquisition QC: Standardized scanning protocols and fixed procedures are used for imaging data acquisition, including the use of specialized earplugs and head fixation pads to reduce noise and motion artifacts. Criteria for data re-acquisition or exclusion are established for subjects with excessive head motion or inability to cooperate.

Data Management: Prospective data collection utilizes unified, standardized questionnaires performed by trained research personnel with simultaneous double verification. All data will be anonymized and stored in an encrypted, dedicated database with strict tiered access control to ensure data security and privacy.

Process and Ethical Oversight: The study protocol, informed consent forms, and other documents have been reviewed and approved by the hospital's Life Ethics Committee. A participant follow-up safeguard mechanism has been established, including follow-up reminders, emergency plans for clinical changes, and documentation of loss to follow-up. The study guarantees participants the right to withdraw unconditionally at any time, with their legitimate rights and interests fully protected.

Sample Size and Statistical Analysis:

The sample size was calculated based on between-group comparisons of the primary outcome measure (MoCA score). Using a one-way ANOVA, with α=0.05, power of 80%, and an effect size f=0.10, the minimum required sample size was calculated to be 1200. Considering a 15% attrition rate, the final planned enrollment is 1500 participants.

Statistical analysis will be performed using SPSS 26.0 and SPM12 software. Continuous data will be described using mean ± standard deviation or median based on normality test results. Between-group comparisons will use ANOVA or non-parametric tests according to data distribution. For multimodal imaging data, voxel-wise between-group comparisons will be conducted, controlling for covariates such as age and sex, with cluster-level FDR correction. Correlation analyses will use Pearson or Spearman correlation, with Bonferroni correction for multiple comparisons. The significance level is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years.
2. Patients clinically diagnosed with CKD stages 1-5.
3. No contraindications for MRI examination (e.g., cardiac pacemaker, claustrophobia, cochlear implant, hearing aid, coronary stents implanted before 2015) and able to complete the MRI scan.

Exclusion Criteria:

1. Patients with recent or prior cerebral hemorrhage or cerebral infarction.
2. History of epileptic seizures or psychiatric disorders.
3. Patients with claustrophobia.
4. Pregnant or lactating patients.
5. Presence of other central nervous system diseases (e.g., tumor, trauma).
6. Unstable angina, congestive heart failure (NYHA class III or IV), or acute myocardial infarction.
7. Any systemic or other diseases deemed unsuitable for clinical trial participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a prospective cohort of adult patients with Chronic Kidney Disease (CKD) recruited from a single clinical center. All participants will be selected from patients attending the Department of Nephrology and other relevant clinics at Beijing Friendship Hospital, Capital Medical University. The primary eligibility criteria include an age range of 18 to 70 years and a clinical diagnosis of CKD at any stage (1 through 5). Key exclusions are applied to ensure patient safety and specificity of the observational findings, primarily concerning conditions that contraindicate MRI procedures or represent significant, unstable comorbid systemic, cardiovascular, or neuropsychiatric diseases. A total of 1500 participants meeting these criteria are planned to be enrolled. Each participant will undergo a comprehensive baseline assessment and a follow-up evaluation at 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function assessed by Montreal Cognitive Assessment (MoCA) | Baseline and 3-year follow-up.
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening tool with a total score range of 0 to 30, where higher scores indicate better cognitive function. A score below 26 is indicative of cognitive impairment.

SECONDARY OUTCOMES:
Retinal Nerve Fiber Layer (RNFL) Thickness | Baseline and 3-year follow-up.
  Thickness of the retinal nerve fiber layer, measured in micrometers (μm) using optical coherence tomography (OCT).
Average Macular Thickness | Baseline and 3-year follow-up.
  The average thickness of the macular region, measured in micrometers (μm) via optical coherence tomography (OCT).
Retinal Specific Lesion Count | Baseline and 3-year follow-up.
  The number of specific lesions (e.g., microaneurysms, hemorrhages) identified in the retina, reported as a count.
Retinal Capillary Plexus Vessel Density (VD) | Baseline and 3-year follow-up.
  The density of blood flow in the retinal capillary networks, expressed as a percentage (%) measured by optical coherence tomography angiography (OCTA).
Retinal Non-Perfusion Area (NPA) | Baseline and 3-year follow-up.
  The total area of retinal capillary non-perfusion, measured in square millimeters (mm²) using optical coherence tomography angiography (OCTA).
Subfoveal Choroidal Thickness (SCT) | Baseline and 3-year follow-up.
  The thickness of the choroid directly beneath the fovea, measured in micrometers (μm) using enhanced-depth imaging optical coherence tomography (EDI-OCT).
Renal Blood Flow (RBF) | Baseline and 3-year follow-up.
  Volume of blood delivered to the kidneys per unit time, measured in milliliters per minute (mL/min).
Estimated Glomerular Filtration Rate (eGFR) | Baseline and 3-year follow-up.
  An estimate of the rate at which blood is filtered by the glomeruli of the kidneys, standardized to body surface area and reported in mL/min/1.73 m².
Albumin | Baseline and 3-year follow-up.
  Concentration of albumin protein in the blood, measured in grams per liter (g/L), important for assessing nutritional status and liver/kidney function.
Hemoglobin (Hb) | Baseline and 3-year follow-up.
  Concentration of hemoglobin in the blood, measured in grams per liter (g/L), indicating the oxygen-carrying capacity of red blood cells.
Uric Acid | Baseline and 3-year follow-up.
  Concentration of uric acid in the blood, measured in micromoles per liter (μmol/L), used as a marker for conditions like gout and kidney function.
Creatinine | Baseline and 3-year follow-up.
  Concentration of creatinine in the blood, measured in micromoles per liter (μmol/L), a key indicator of kidney function.
High-sensitivity C-Reactive Protein (hs-CRP) | Baseline and 3-year follow-up.
  Concentration of albumin protein in the blood, measured in grams per liter (g/L), important for assessing nutritional status and liver/kidney function.
Serum Phosphate | Baseline and 3-year follow-up.
  Concentration of inorganic phosphate in the blood, measured in millimoles per liter (mmol/L), important for bone metabolism and cellular energy.
Serum Calcium | Baseline and 3-year follow-up.
  Concentration of calcium in the blood, measured in millimoles per liter (mmol/L), crucial for bone health, nerve function, and blood clotting.
Gray Matter Volume (GMV) | Baseline and 3-year follow-up.
  The volume of gray matter tissue in a specific region of the brain, measured in cubic millimeters (mm³) from structural magnetic resonance imaging (MRI).
Amplitude of Low-Frequency Fluctuations (ALFF) | Baseline and 3-year follow-up.
  A measure of the intensity of regional spontaneous brain activity in the low-frequency range, derived from resting-state functional MRI (fMRI) and expressed in arbitrary units (a.u.).
Cerebral Blood Flow (CBF) | Baseline and 3-year follow-up.
  The volume of blood supplying a given amount of brain tissue per unit time, typically measured in milliliters per 100 grams of tissue per minute (mL/100 g/min) using arterial spin labeling (ASL) or similar MRI techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided